CLINICAL TRIAL: NCT06794736
Title: STRatifying Adult DIffuse Lower-grade Gliomas Based on Their VARIed Metabolic Profiles (STRADIVARI Project)
Acronym: STRADIVARI
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Collaborators: Università Vita-Salute San Raffaele (Other); University of Bari (Other); Ospedale San Paolo Bari (Unknown)
Responsible Party: Sponsor
Other Study IDs: STRADIVARI
Record Dates: First submitted 2025-01-15; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Lower Grade Glioma
Keywords: Lower grade glioma; Metabolomics; Tumor heterogeneity; Patient Stratification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Fresh glioma samples from prospective cohort FFPE section from retrospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective Metabolic Cohort: Patients operated on for lower grade gliomas from whom part of the exceeding pathologic material will be collected for metabolomic profiling
- Retrospective FFPE Sample Cohort: Historical patient cohort for whom FFPE sections, full clinical history and pathological data are available.

SUMMARY:
The goal of this observational study is to better characterise lower-grade gliomas from a molecular and metabolic point of view, so to identify further subgroups of these tumours with different behaviour and, possibly, different treatment susceptibility.

Participants of prospective metabolic cohort will be subjected to routine treatment, part of the exceeding tutor material will be subjected to advanced molecular-metabolic analyses to desume their metabolic profile to be then correlated with clinical outcome (progression-free survival, overall survival, response to therapy/progression) and diagnosis (astrocytoma/oligodendroglioma and grade).

Critical enzymes identified from metabolic analyses on the first cohort will be tested on a protein level on a retrospective cohort of patients previously operated and for whom fully available clinical history and pathological material is available in Institutional archive (no need for further intervention on these patients) to see if they actually correlate with clinical outcome.

ELIGIBILITY:
Prospective Metabolic Cohort:

Inclusion Criteria:

* Radiological diagnosis of brain tumor compatible with lower grade glioma
* Full clinical history

Exclusion Criteria:

* Current pregnancy or lactation
* Patients not able to provide informed consent

Retrospective Cohort of FFPE samples:

Inclusion Criteria:

* Confirmed diagnosis of lower grade glioma
* Full clinical and radiological history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by brain lower grade gliomas who access Neurosurgery Department (OR, ER, outpatient clinic) at IRCCS Ospedale Galeazzi Sant'Ambrogio and Policlinico Bari, or Oncology Department at Ospedale San Paolo Bari
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | (up to 180 months)
  time from surgery to evidence of radiological progression at MRI
Overall Survival (OS) | (up to 180 months)
  Time from surgery to tumor-related death

SECONDARY OUTCOMES:
Histological-molecular diagnosis (integration of immunohistochemistry and molecular evaluation of IDH1/2, ATRX and 1p/19q chromosomal deletion) | From date of surgery to date of complete diagnosis (weeks)
  Astrocytoma vs Oligodendroglioma (integration of immunohistochemistry and molecular evaluation of IDH1/2, ATRX and 1p/19q chromosomal deletion)
Tumor Grade at histology and molecular analysis (CDKN2A/B deletion) | From surgery to complete history-molecular diagnosis (weeks)
  Tumor grade upon histology and molecular analysis (CDKN2A/B deletion)

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Ospedale San Paolo Bari, Bari, Apulia
  - Policlinico Bari University Hospital (Bari, Italy), Bari, Apulia
  - Università Vita-Salute San Raffaele, Milan, Lombardy
  - IRCCS Galeazzi-Sant'Ambrogio, Milan, Lombardy

IPD SHARING:
Plan to Share IPD: Undecided